CLINICAL TRIAL: NCT00144599
Title: A Double-Blind, Phase III Study to Evaluate the Efficacy, Safety and PK of MRA in Patients With sJIA
Brief Title: Study of MRA for Systemic Juvenile Idiopathic Arthritis (sJIA)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chugai Pharmaceutical (Industry)
Responsible Party: Chugai Pharmaceutical, Chugai Pharmaceutical
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MRA316JP
Record Dates: First submitted 2005-09-02; First posted 2005-09-05 (Estimated); Last update posted 2008-07-30 (Estimated); Status verified 2008-07

CONDITIONS: Systemic Juvenile Idiopathic Arthritis
MeSH Terms: conditions — Arthritis, Juvenile | interventions — tocilizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: MRA(Tocilizumab)
- 2 (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: MRA(Tocilizumab)
  Arms: 1
Drug: placebo
  Arms: 2

SUMMARY:
This is a double-blind, Phase III study to evaluate the efficacy, safety and PK of MRA in patients with sJIA.

ELIGIBILITY:
Inclusion criteria

* Patients diagnosed as having systemic JIA based on the International League of Associations for Rheumatology criteria (1997)
* Patients between 2 and 19 years of age
* Patients who are under 16 years of age at onset
* Patients who have been treated with corticosteroids (continued treatment for 3 months or longer at a dose of ≥0.2 mg/kg as prednisolone equivalent) but who failed to respond adequately or in whom treatment could not be continued or the dose could not be increased due to adverse drug reactions

Exclusion criteria

* Patients who have been treated with infliximab or etanercept within 12 weeks before treatment with the investigational product
* Patients who have received the following treatments within 4 weeks before treatment with the investigational product

  1. Surgical treatment (e.g., operation)
  2. Plasma exchange therapy"

Ages: 2 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 56 (Actual)
Dates: Start 2004-05; Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
Efficacy:Percentage of patients showing 30% improvement in the JIA core set, Percentage of patients showing improvement in CRP on LOBS | open-label period
Efficacy:Percentage of patients in whom effects were maintained | Blind period
Safety:Incidence and severity of adverse events and adverse drug reactions | whole period
Pharmacokinetics:The time course of the trough serum MRA concentration | whole period

SECONDARY OUTCOMES:
Efficacy:Time courses of CRP and ESR, percentage of patients showing 30%, 50%, and 70% improvement in the JIA core set, JIA core set variables, pain, maximum body temperature, systemic feature score | Open-label period
Period for which effects, Time course of CRP and ESR, percentage of patients showing 30%, 50%, and 70% improvement in the JIA core set,JIA core set variables,pain, maximum body temperature,systemic feature score up to LOBS | Blind Period

CONTACTS AND LOCATIONS:
Overall Officials: Takahiro Kakehi, Study Director — Chugai Pharmaceutical

REFERENCES:
- [Derived] Aoki C, Inaba Y, Choe H, Kaneko U, Hara R, Miyamae T, Imagawa T, Mori M, Oba MS, Yokota S, Saito T. Discrepancy between clinical and radiological responses to tocilizumab treatment in patients with systemic-onset juvenile idiopathic arthritis. J Rheumatol. 2014 Jun;41(6):1171-7. doi: 10.3899/jrheum.130924. Epub 2014 May 1. PMID 24786929
- [Derived] Yokota S, Imagawa T, Mori M, Miyamae T, Takei S, Iwata N, Umebayashi H, Murata T, Miyoshi M, Tomiita M, Nishimoto N, Kishimoto T. Longterm safety and effectiveness of the anti-interleukin 6 receptor monoclonal antibody tocilizumab in patients with systemic juvenile idiopathic arthritis in Japan. J Rheumatol. 2014 Apr;41(4):759-67. doi: 10.3899/jrheum.130690. Epub 2014 Mar 15. PMID 24634205
- [Derived] Yokota S, Imagawa T, Mori M, Miyamae T, Aihara Y, Takei S, Iwata N, Umebayashi H, Murata T, Miyoshi M, Tomiita M, Nishimoto N, Kishimoto T. Efficacy and safety of tocilizumab in patients with systemic-onset juvenile idiopathic arthritis: a randomised, double-blind, placebo-controlled, withdrawal phase III trial. Lancet. 2008 Mar 22;371(9617):998-1006. doi: 10.1016/S0140-6736(08)60454-7. PMID 18358927